CLINICAL TRIAL: NCT00492297
Title: A Phase II, Multi-center, Open-label, Uncontrolled Study to Evaluate the Efficacy and Safety of BAY 43-9006 Given Daily in Combination With Repeated 21-Day Cycles of Dacarbazine (DTIC) Chemotherapy in Subjects With Advanced Metastatic Melanoma.
Brief Title: A Phase II, Multi-Center, Open-Label, Uncontrolled Study to Evaluate the Efficacy and Safety of Sorafenib Given Daily in Combination With Repeated 21-Day Cycles of Dacarbazine (DTIC) Chemotherapy in Subjects With Advanced Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11538; 2004-000725-30 (EudraCT Number)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib + Dacarbazine (Experimental): Dacarbazine 1000 mg/m^2 on day one of repeated 21 day cycles, in combination with daily continuous oral sorafenib (Nexavar, BAY 43-9006), 400 mg twice a day (bid)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine (DTIC)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine (DTIC) — Dacarbazine 1000 mg/m^2 on day one of repeated 21 day cycles, in combination with daily continuous oral sorafenib (Nexavar, BAY 43-9006), 400 mg twice a day (bid)

SUMMARY:
The purpose of this study is to see whether a new type of anti-cancer drug, known as BAY 43-9006, can be given safely and with good effect in combination with dacarbazine (DTIC). DTIC is the current standard chemotherapy drug given for melanoma that has spread through the body. Although this drug can be effective on its own and is generally well tolerated, not all patients will benefit, so there is a need to test new drugs and drug combinations for treating melanoma.

DETAILED DESCRIPTION:
Issues on "Safety" outcomes are addressed in the Adverse Event section.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced, metastatic, histologically confirmed melanoma, for whom treatment with dacarbazine is considered medically acceptable
* Age >= 18 years
* Subject has measurable and evaluable disease defined as at least one metastatic lesion that can be accurately and serially measured by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scan as per the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Cutaneous lesions measuring at least 20mm in longest diameter can be considered measurable (and therefore target lesions) via color photography including a ruler
* Subject has biopsiable disease at baseline and is willing to provide biopsy samples, or does not have biopsiable disease at baseline
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Primary ocular or mucosal melanoma (cutaneous vulval melanoma is permitted)
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry
* (Active coronary artery disease or ischemia (myocardial infarction more than 6 months prior to study entry is allowed)
* Uncontrolled hypertension (> grade 2 National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0)
* Active, clinically serious infections (> grade 2 NCI-CTCAE version 3.0)
* Subjects with seizure disorder requiring medication are excluded
* History of or suspected Human Immunodeficiency Virus (HIV) infection, or chronic hepatitis B or C
* Symptomatic metastatic brain or meningeal tumors unless the subject is > 6 months from definitive therapy, has a negative imaging study within 4 weeks prior to study entry and is clinically stable with respect to the tumor at the time of study entry. Also the subject must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies)
* Pregnant or breast-feeding subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- France (4):
  - Bordeaux
  - Lyon
  - Toulouse
  - Villejuif
- United Kingdom (6):
  - Cambridge, Cambridgeshire
  - Southampton, Hampshire
  - London, London
  - Manchester, Manchester
  - Northwood, Middlesex
  - Sutton, Surrey

REFERENCES:
- [Result] Eisen T, Marais R, Affolter A, Lorigan P, Robert C, Corrie P, Ottensmeier C, Chevreau C, Chao D, Nathan PD, Jouary T, Harries M, Negrier S, Montegriffo E, Ahmad T, Gibbens I, James MG, Strauss UP, Prendergast S, Gore ME. Sorafenib and dacarbazine as first-line therapy for advanced melanoma: phase I and open-label phase II studies. Br J Cancer. 2011 Jul 26;105(3):353-9. doi: 10.1038/bjc.2011.257. Epub 2011 Jul 12. PMID 21750549
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had a 2-stage Simon optimal design consisting of 30 subjects in the first stage and 52 subjects in the second stage for a planned total of 82 subjects. Actually a total of 96 subjects were enrolled and 83 were treated; 32 in the 1st stage and 51 in the second stage. The study was conducted at 8 centers in the UK and 4 centers in France.
Pre-assignment Details: Of the 96 enrolled subjects, 13 were screening failures. The reasons for screening failure were violation of inclusion/exclusion criteria (12) and death due to Progressive Disease (PD) (1). The remaining 83 subjects all received at least one dose of sorafenib and dacarbazine.
Groups:
- Sorafenib + Dacarbazine: Dacarbazine 1000 mg/m^2 on day one of repeated 21 day cycles, in combination with daily continuous oral Sorafenib (Nexavar, BAY43-9006), 400 mg twice a day (bid), the treatment continued until subjects had clear palliative benefit and were tolerating treatment well, or until progressive disease (PD) or death (if earlier) recorded up to 97 weeks. Subjects withdrawn from Sorafenib but with optional standard treatment entered Active Follow-up (AFU) period, which was 30(+4) days for subjects who had PD at the end of treatment; or until PD was documented for subjects who had complete response (CR) or partial response (PR) or stable disease (SD) at the end of treatment up to 97 weeks . Once subject progressed went into survival only follow-up which continued until death occurred up to 172 weeks.
Period: Treatment
Arm/Group | Sorafenib + Dacarbazine
Started | 83
First Stage of Simon Optimal Design | 32 (32 subjects of 83 subjects enrolled were treated in first stage.)
Second Stage of Simon Optimal Design | 51 (Recruitment continued into the second stage. 51 of 83 subjects were treated in the second stage.)
Completed | 78
Not Completed | 5
Not completed — Death | 2
Not completed — Study terminated by sponsor | 3
Period: Active Follow-up 30(+4) Days Duration
Arm/Group | Sorafenib + Dacarbazine
Started | 78 (AFU is 30(+4) days duration for subjects withdrawn from sorafenib due to PD.)
Completed | 59
Not Completed | 19
Not completed — Death | 17
Not completed — Study terminated by sponsor | 2
Period: Survival Only Follow-up
Arm/Group | Sorafenib + Dacarbazine
Started | 59
Completed | 0
Not Completed | 59
Not completed — Death | 46
Not completed — Lack of Efficacy | 1
Not completed — Study terminated by sponsor | 12

BASELINE CHARACTERISTICS:
Groups:
- Sorafenib + Dacarbazine: Dacarbazine 1000 mg/m2 on day one of repeated 21 day cycles, in combination with daily continuous oral Sorafenib (Nexavar, BAY43-9006), 400 mg twice a day (bid)
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 83
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [25 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 50
Clinical disease status [Number; unit: participants] — Clinical disease status at the beginning of the study. Stable Disease (SD): No change in tumor size. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since treatment started, or the appearance of 1 or more new lesions.
  participants
    Missing | 6
    Stable disease | 3
    Progressive disease | 74
Disease stage (AJCC) [Number; unit: participants] — Disease stage according to the American Joint Committee on Cancer (AJCC) based on the TNM (tumor-node-metastasis) classification. Stage I and stage II (T2bN0M0-T4bN0M0) is localized disease, stage III (Any T1-4a, N1bM0-AnyTN3M0) is locally advanced disease and stage IV (Any T, Any N, Any M except M0) is metastatic disease.
  participants
    Missing | 1
    M1a Distant subcutaneous or lymphnode metastases | 4
    M1b Lung metastases | 12
    M1c All other visceral metastases | 66
ECOG status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects a patient. The scale ranges from 0 (fully active) to 5 (dead). Subjects entering this study must have had an ECOG score of 0 or 1 (restricted in physically strenuous activity but ambulatory).
  participants
    Missing | 3
    0 | 52
    1 | 28
Histology [Number; unit: participants] — Histologically confirmed melanoma was one of the inclusion criteria for enrollment into the study. This information was collected at the time of enrollment and included in the patient's record.
  participants
    Missing | 24
    Malignant melanoma | 4
    Superfical spreading | 24
    Nodular | 29
    Acral lentiginous | 2
Lactate dehydrogenase [Number; unit: participants] — Tissue breakdown elevates levels of lactate dehydrogenase (LDH). LDH can be elevated in several disorders, including cancer.
  participants
    Missing | 3
    < Upper Limit of Normal (ULN=325 U/L) | 43
    >= ULN but < 10 percent above ULN | 11
    >= 10 percent above the ULN | 26
Mean time from diagnosis [Mean (Full Range); unit: days] — Mean number of days from initial diagnosis to randomization into the study.
  days | 1280 [9 to 5344]

OUTCOME MEASURES:

1. Primary Outcome: Overall Best Response
Description: Best Overall Response (BOR): Best tumor response achieved during or within 30 days after active therapy confirmed according to the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR): The disappearance of all target and non-target lesions. Partial response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. SD was defined as steady state of disease, PD was defined as an increase of at least 20% increase in the sum of the LD of target lesions or appearance of new lesions.
Time Frame: during or within 30 days after active therapy
Population: There were 83 subjects in the intent-to-treat (ITT) population. Of these, 75 were evaluable for Best Response; 8 were not evaluable.
Measure: Number; unit: participants
Groups:
- Sorafenib + Dacarbazine: Dacarbazine 1000 mg/m^2 on day one of repeated 21 day cycles, in combination with daily continuous oral Sorafenib (Nexavar, BAY43-9006), 400 mg twice a day (bid)
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 75
participants
  Overall response (CR+PR) | 10
  Complete response (CR) | 1
  Partial response (PR) | 9
  Stable disease (SD) | 31
  Progressive disease (PD) | 34

2. Secondary Outcome: Progression-free Survival
Description: Progression-free Survival (PFS) was the time from the first dose of combination therapy to disease progression (radiological or clinical, whichever is earlier) or death (if death occurs before progression is documented). PFS for subjects without tumor progression or death at the time of analysis were censored at the date of last tumor evaluation.
Time Frame: from start of treatment until progression or death before progression (median 259 days)
Population: There were 83 subjects in the intent-to-treat (ITT) population. All 83 were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 83
days | 102 [83 to 134]

3. Secondary Outcome: Percentage of Subjects With Progression-free Survival at Specific Time-points
Description: as for outcome 2
Time Frame: from start of treatment until progression or death before progression after 3, 6 and 12 months
Population: There were 83 subjects in the intent-to-treat (ITT) population. All 83 were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 83
percentage of participants
  PFS at month 3 | 56.63
  PFS at month 6 | 33.73
  PFS at month 12 | 10.84

4. Secondary Outcome: Overall Survival
Description: Overall Survival was the number of days from the date that combination treatment started until the date of death.
Time Frame: from start of treatment until death (median 259 days)
Population: There were 83 subjects in the intent-to-treat (ITT) population. All 83 were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 83
days | 259 [237 to 322]

5. Secondary Outcome: Duration of Response
Description: Duration of Response was assessed in subjects who showed a Partial Response (PR) or Complete Response (CR). It was defined as the time from the first documented objective response to Progressive Disease (PD), or death if before documented progression. Duration of response for subjects who have not progressed or died at the time of analysis was censored at the date of last tumor assessment.
Time Frame: from confirmed Complete Response (CR) or Partial Response (PR) until Progressive Disease (PD) (median 259 days)
Population: There were 83 subjects in the intent-to-treat (ITT) population. Only the 10 subjects who had a PR or CR were included in this analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 10
days | 327 [99 to 628]

6. Secondary Outcome: Duration of Complete Response
Description: Duration of complete response was the number of days from the date that a complete response was first documented to the date that recurrent or progressive disease was first objectively documented (if patient progressed then censored=no) or to last observation (if patient did not progress then censored=yes).
Time Frame: from confirmed CR until PD (median 259 days)
Population: There were 83 subjects in the intent-to-treat (ITT) population. Only the 1 subject who had a CR was included in this analysis (duration 420 days, censored).
Measure: Number; unit: days
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 1
days | 420

7. Secondary Outcome: Duration of Partial Response
Description: Duration of partial response was the number of days from the date that a partial response was first documented to the date that recurrent or progressive disease was first objectively documented (if patient progressed then censored=no) or to last observation (if patient did not progress then censored=yes).
Time Frame: from confirmed PR until PD (median 259 days)
Population: There were 83 subjects in the intent-to-treat (ITT) population. Only the 9 subjects who had a PR were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 9
days | 255 [231 to 448]

8. Secondary Outcome: Disease Control (DC)
Description: DC was defined as the total number of subjects whose best response was not progressive disease (PD) (total number of CRs + total number of PRs + total number of Stable Diseases (SD)). The DC at specific time points could also be calculated as the total number of subjects whose response was not PD at that time point.
Time Frame: after start of treatment, at 6 months and 12 months
Population: There were 83 subjects in the intent-to-treat (ITT) population. All 83 were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 83
participants
  DC based on overall best response | 41
  DC at 6 months | 38
  DC at 12 months | 38

9. Secondary Outcome: Duration of Stable Disease
Description: Duration of Stable Disease (DSD), defined as the time from the first documented objective evidence of Stable Disease (SD) to disease progression (DP) or death if death occurred before DP, was assessed in subjects who showed SD as best response. DSD for subjects who had not progressed or died was censored at the date of last tumor assessment.
Time Frame: from start of therapy to PD, only in non-responders (median 259 days)
Population: There were 83 subjects in the intent-to-treat (ITT) population. Only the 70 subjects who had a Best Response of Stable Disease, ie, those who failed to achieve a Best Response of CR or PR, were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 70
days | 93 [77 to 112]

10. Secondary Outcome: Time to Response
Description: Time to Response in subjects who achieved an objective response (PR or CR with confirmation) was measured from the date of starting study combination treatment until the earliest date that the response was first documented.
Time Frame: start of therapy to confirmed CR or PR (median 259 days)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 10
days | 48 [41 to 87]

11. Secondary Outcome: Time to Progression
Description: Time to Progression was the number of days from the start of therapy to progression (if patient progressed then censored=no) or to the last observation at which the patient was known to have not progressed, that is, the last observation with a best response of CR, PR, or SD.
Time Frame: From start of treatment until progression (median 259 days)
Population: There were 83 subjects in the intent-to-treat (ITT) population. Of these 83, 78 were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Dacarbazine
Number analyzed (Participants) | 78
days | 102 [88 to 139]

ADVERSE EVENTS:
Description: The following abbreviations were used in the Adverse Event section: - Q-T Corrected (QTc) - Common Terminology Criteria for Adverse Events (CTCAE) - Not Otherwise Specified (NOS) - Gastrointestinal (GI) - Alanine aminotransferase (ALT)
Arm/Group | Sorafenib + Dacarbazine
Serious Adverse Events (participants affected / at risk) | 40/83
Other Adverse Events (participants affected / at risk) | 82/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Dacarbazine (N=83)
Blood - other (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 3
Leukocytes (Blood and lymphatic system disorders) | 2
Neutrophile (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 5
Cardiac arrhythmia - other (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Prolonged QTC (Cardiac disorders) | 1
Supraventricular arrhythmia, atrial fibrillation (Cardiac disorders) | 2
Cardiac ischemia/infarction (Cardiac disorders) | 2
Fatigue (General disorders) | 3
Fever (General disorders) | 4
Death not associated with CTAE term, disease progression nos (General disorders) | 7
Dermatology - other (Skin and subcutaneous tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hemorrhage - other (Vascular disorders) | 1
Hemorrhage, GI, lower GI (Vascular disorders) | 1
Hemorrhage, GI, upper GI nos (Vascular disorders) | 1
Hepathobiliary - other (Hepatobiliary disorders) | 1
Liver dysfunction (Hepatobiliary disorders) | 1
Febrile neutropenia (Infections and infestations) | 1
Infection (doc. clinic), foreign body (e.g. graft, implant, pros, stent) (Infections and infestations) | 1
Infection (documented clinically), lung (pneumonia) (Infections and infestations) | 1
Infection (documented clinically), upper airway nos (Infections and infestations) | 1
Infection - other (Infections and infestations) | 2
Device/prosthesis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Neurology - other (Nervous system disorders) | 1
Ocular - other (Eye disorders) | 1
Pain, abdomen nos (General disorders) | 5
Pain, chest/thorax nos (General disorders) | 2
Pain, head/headache (General disorders) | 2
Pain, other (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Renal - other (Renal and urinary disorders) | 1
Secondary malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Dacarbazine (N=83)
Neutrophils (Blood and lymphatic system disorders) | 42
Hemoglobin (Blood and lymphatic system disorders) | 15
Platelets (Blood and lymphatic system disorders) | 24
Leukocytes (Blood and lymphatic system disorders) | 15
Cardiac arrhythmia - other (Cardiac disorders) | 5
Hypertension (Cardiac disorders) | 16
Fever (General disorders) | 10
Fatigue (General disorders) | 51
Constitutional symptoms - other (General disorders) | 7
Sweating (General disorders) | 10
Anorexia (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 44
Diarrhea (Gastrointestinal disorders) | 43
Gastritis (Gastrointestinal disorders) | 5
Heartburn (Gastrointestinal disorders) | 8
Mucositis (functional/symptomatic), oral cavity (Gastrointestinal disorders) | 6
Mucositis (clinical exam), oral cavity (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 38
Vomiting (Gastrointestinal disorders) | 24
Infection - other (Infections and infestations) | 13
ALT (Metabolism and nutrition disorders) | 5
Amylase (Metabolism and nutrition disorders) | 5
Metabolic/lab - other (Metabolism and nutrition disorders) | 6
Mood alteration, depression (Nervous system disorders) | 6
Neurology - other (Nervous system disorders) | 7
Neuropathy: Sensory (Nervous system disorders) | 19
Pain, back (General disorders) | 10
Pain, chest/thorax nos (General disorders) | 5
Pain, extremity-limb (General disorders) | 14
Pain, abdomen nos (General disorders) | 24
Pain, head/headache (General disorders) | 16
Pain, joint (General disorders) | 16
Pain, other (General disorders) | 7
Pain, pelvis (General disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10
Voice changes (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 20
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 37
Dermatology - other (Skin and subcutaneous tissue disorders) | 22
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 33
Flushing (Skin and subcutaneous tissue disorders) | 16

LIMITATIONS AND CAVEATS:
Due to the small number of patients, no conclusions can be drawn from these data in terms of BRAF mutations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication will be discussed with the sponsor prior to release and written consent of the sponsor will be obtained. A draft manuscript of the publication or abstract must be sent to sponsor thirty days in advance of submission.